CLINICAL TRIAL: NCT05525689
Title: Technology-Enabled Services to Support Care Mangers in Obstetrics Clinics to Treat Perinatal Depression
Brief Title: Evaluating Technology Enabled Services in Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Brown University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Mohr, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH119029-RP2-RCT; 5P50MH119029-04 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-09-01 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Perinatal
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Enabled Service (Experimental): Access to the Intellicare suite of digital mental health self-management tools and coaching
  Interventions: Behavioral: IntelliCare
- eTreatment as Usual (Active Comparator): Current care plus access to a website that will provide content specific to perinatal depression
  Interventions: Other: COMPASS-Care

INTERVENTIONS:
Behavioral: IntelliCare — Application with patient-facing tools for depression symptom monitoring, self-management, and care manager communication as well as care manager dashboards for workflow optimization
  Arms: Technology Enabled Service
Other: COMPASS-Care — Website with content specific to perinatal depression and standard EHR-based tools for patient communication
  Arms: eTreatment as Usual

SUMMARY:
Investigators are evaluating a Technology Enabled Service (TES) to support the treatment of depression in the context of a collaborative care service in obstetrics clinics.

DETAILED DESCRIPTION:
Investigators are evaluating a Technology Enabled Service (TES) to support the treatment of depression in the context of a collaborative care service in obstetrics clinics. The TES consists of digital technologies that connect patients to care managers remotely, providing tools for monitoring patient symptoms, communication, and delivery of a digital intervention. The intervention consists of a patient-facing app for assessment and self-management of depression.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 years or older
* Referred to Northwestern Medicine COMPASS program for mental health care
* Currently pregnant or within 3 months of delivery
* Moderate to severe perinatal depression (defined as a PHQ-9 screen greater than or equal to 10)
* Owns a smartphone, has used smartphone in last 7 days

Exclusion Criteria:

* Experienced a pregnancy loss (miscarriage, termination, or stillbirth of the index pregnancy)
* Severe suicidality (as defined by the presence of a plan and intent to act on that plan)
* Not meeting the inclusion criteria described above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mohr, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Technology Enabled Service | eTreatment as Usual
Started | 38 | 37
Completed | 37 | 37
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Technology Enabled Service | eTreatment as Usual | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 32.0 [28.8 to 35.5] | 33.2 [29.6 to 36.7] | 32.0 [28.8 to 35.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 5 | 22
  White | 13 | 20 | 33
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75
General Health [Count of Participants; unit: Participants]
  Poor | 0 | 1 | 1
  Fair | 8 | 6 | 14
  Good | 16 | 15 | 31
  Very Good | 13 | 14 | 27
  Excellent | 1 | 1 | 2
Engaged in Psychotherapy [Count of Participants; unit: Participants]
  Yes | 23 | 31 | 54
  No | 15 | 6 | 21
Using Psychiatric Medications [Count of Participants; unit: Participants]
  Yes | 13 | 18 | 31
  No | 25 | 19 | 44
Education [Count of Participants; unit: Participants]
  Some high school or less | 1 | 0 | 1
  High School Graduate/ GED | 8 | 4 | 12
  Associate degree | 1 | 1 | 2
  Some college | 11 | 11 | 22
  Bachelor's Degree | 9 | 7 | 16
  Post-bachelor's Education | 8 | 14 | 22
Employed [Count of Participants; unit: Participants]
  Yes | 24 | 28 | 52
  No | 12 | 9 | 21
  Prefer not to answer | 2 | 0 | 2
Income [Count of Participants; unit: Participants]
  Less than $10,000 | 9 | 0 | 9
  $10,000 - $19,999 | 3 | 3 | 6
  $20,000 - $39,999 | 4 | 4 | 8
  $40,000 - $59,999 | 5 | 3 | 8
  $60,000 - $99,999 | 4 | 4 | 8
  $100,000 + | 12 | 19 | 31
  Don't know | 1 | 1 | 2
  Prefer not to answer | 0 | 3 | 3
Marital Status [Count of Participants; unit: Participants]
  Divorced | 1 | 0 | 1
  Domestic partnership | 1 | 1 | 2
  Living with partner | 6 | 6 | 12
  Married | 17 | 25 | 42
  Separated | 1 | 0 | 1
  Single; never married | 12 | 5 | 17
Household Size [Count of Participants; unit: Participants]
  1 | 2 | 0 | 2
  2 | 10 | 10 | 20
  3 | 10 | 18 | 28
  4+ | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Assessed by Patient Health Questionnaire-9
  Scores range from 0-27. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: At 12 weeks
Population: Analysis from all observed data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Technology Enabled Service | eTreatment as Usual
Number analyzed (Participants) | 38 | 37
score on a scale | 6.42 [4.80 to 8.03] | 6.55 [4.90 to 8.20]

2. Secondary Outcome: Anxiety
Description: Assessed by General Anxiety Disorder - 7
  Scores range from 0-21. The following cut-offs correlate with level of anxiety severity:
  Score 0-4: Minimal Anxiety Score 5-9: Mild Anxiety Score 10-14: Moderate Anxiety Score greater than 15: Severe Anxiety
Time Frame: At 12 weeks
Population: From all observed data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Technology Enabled Service | eTreatment as Usual
Number analyzed (Participants) | 38 | 37
score on a scale | 6.57 [5.02 to 8.12] | 7.38 [5.79 to 8.97]

3. Secondary Outcome: Satisfaction Index - Mental Health
Description: The Satisfaction Index - Mental Health measures satisfaction with mental health treatment. The measure includes 12 items, each rated on a 1-6 point likert scale (range of 6-72 points for total score) where higher scores reflect higher satisfaction.
  Scores were analyzed as discrete outcomes at 6 and 12 weeks. Separate analyses were conducted for each time point using the Welch two-sample t-test to compare scores across intervention groups.
Time Frame: Week 6, Week 12
Population: From all observed data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Technology Enabled Service | eTreatment as Usual
Number analyzed (Participants) | 38 | 37
score on a scale
  Week 6 | 58 [47 to 68] | 62 [50 to 67]
  Week 12 | 62 [47 to 68] | 60 [52 to 66]

4. Other Pre Specified Outcome: TWente Engagement With Ehealth Technologies Scale (TWEETS)
Description: The TWEETs measures engagement, usability, usefulness, and satisfaction with the digital mental health tool. It includes 9 items rated on 1-5 point likert scales, and produces a total score ranging from 9 to 45. Higher scores indicate better usability.
  TWEETS scores were analyzed as discrete outcomes at 6 and 12 weeks. Separate analyses were conducted for each time point using the Welch two-sample t-test to compare scores across intervention groups.
Time Frame: Week 6, Week 12
Population: from all observed data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Technology Enabled Service | eTreatment as Usual
Number analyzed (Participants) | 38 | 37
score on a scale
  Week 6 | 38 [30 to 43] | 26 [22 to 32]
  Week 12 | 35 [28 to 42] | 27 [24 to 36]

5. Other Pre Specified Outcome: Execution of Stepped Care
Description: Proportion of eligible women engaged in stepped care treatment (# of women who got stepped care / # of women in whom it was indicated (i.e., PHQ9 >=10))
Time Frame: Up to 12 weeks
Population: Analysis only completed on patients meeting criteria for stepped care, as described.
Measure: Count of Participants; unit: Participants
Arm/Group | Technology Enabled Service | eTreatment as Usual
Number analyzed (Participants) | 19 | 10
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored throughout participant involvement in the clinical trial, up to 12 weeks.
Arm/Group | Technology Enabled Service | eTreatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT05525689/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT05525689/SAP_001.pdf
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05525689/ICF_002.pdf